CLINICAL TRIAL: NCT00802360
Title: A Multi-Center, Randomized, Open-Label Evaluation of MENOPUR® Versus FOLLISTIM® in GnRH Antagonist Cycles
Brief Title: MENOPUR® Versus FOLLISTIM®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-04
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Infertility
Keywords: Healthy, pre-menopausal women, age 18-42 with a history of infertility and requiring IVF
MeSH Terms: conditions — Infertility | interventions — Menotropins; Progesterone; follitropin beta; Oils; ganirelix; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Menopur/Endometrin (Experimental): Highly purified menotropin (Menopur®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progestrone vaginal insert (Endometrin®) starts on the day following oocyte retrieval and continues for a total duration of 10 weeks or until a negative pregnancy test is obtained.
  Interventions: Drug: Menotropin; Drug: Progestrone vaginal insert; Drug: Ganirelix
- Menopur/Progesterone in Oil (Experimental): Highly purified menotropin (Menopur®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone in Oil injections start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
  Interventions: Drug: Menotropin; Drug: Progesterone in oil; Drug: Ganirelix
- Follistim/Endometrin (Active Comparator): Follitropin beta (Follistim®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progestrone vaginal insert (Endometrin®) starts on the day following oocyte retrieval and continues for a total duration of 10 weeks or until a negative pregnancy test is obtained.
  Interventions: Drug: Progestrone vaginal insert; Drug: follitropin beta; Drug: Ganirelix
- Follistim/Progesterone in Oil (Active Comparator): Follitropin beta (Follistim®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone in Oil injections start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
  Interventions: Drug: follitropin beta; Drug: Progesterone in oil; Drug: Ganirelix

INTERVENTIONS:
Drug: Menotropin — 225 IU (up to 450 IU) by subcutaneous injection once per day for up to about 15 days until human chorionic gonadotropin (hCG) criteria are met.
  Other Names: highly purified menotropins; Menopur®; hMG
  Arms: Menopur/Endometrin; Menopur/Progesterone in Oil
Drug: Progestrone vaginal insert — 100 mg progesterone vaginal insert 2 or 3 times daily (BID or TID) (start on the day after oocyte retrieval) until 10 weeks gestation or confirmation of negative pregnancy test.
  Other Names: progesterone; Endometrin®
  Arms: Follistim/Endometrin; Menopur/Endometrin
Drug: follitropin beta — 225 IU (up to 450 IU) by subcutaneous injection once per day for up to about 15 days until human chorionic gonadotropin (hCG) criteria are met.
  Other Names: Follistim Pen®; Follistim®
  Arms: Follistim/Endometrin; Follistim/Progesterone in Oil
Drug: Progesterone in oil — 50 mg by intramuscular injection once per day, starting on the day after oocyte retrieval until 10 weeks gestation or confirmation of negative pregnancy test.
  Arms: Follistim/Progesterone in Oil; Menopur/Progesterone in Oil
Drug: Ganirelix — Ganirelix acetate 250 µg as a daily subcutaneous injection starting on day 6 and continuing until hCG criteria were met.
  Other Names: ganirelix acetate; GnRH antagonist

SUMMARY:
To compare the efficacy and safety of highly purified menotropin (Menopur®) with that of follitropin beta (FOLLISTIM®) in patients who are undergoing gonadotropin-releasing hormone (GnRH) antagonist in vitro fertilization (IVF) cycles

DETAILED DESCRIPTION:
This multicenter, randomized, open-label exploratory study will be performed in approximately 200 healthy females undergoing in vitro fertilization (IVF). Each study center will follow its study center standard practice for in vitro fertilization (IVF) within the study parameters as noted in this protocol. The study centers will use marketed products purchased from Schraft's Pharmacy for all phases of the study (down-regulation, stimulation, ovulation induction, and luteal support). Subjects will be randomly assigned prior to the start of stimulation to highly purified menotropin (Menopur®) or follitropin beta (Follistim Pen®) for stimulation and progesterone vaginal insert (Endometrin®) or progesterone in oil for luteal support. Subjects will return to the study center for regular scheduled clinic visits as required per in vitro fertilization (IVF) protocol at the site and at specified time periods during the cycle for estradiol (E2), progesterone (P4) and human chorionic gonadotropin (hCG) tests, and first serum pregnancy test. All subjects will be required to complete a final study visit at completion of luteal support or negative serum pregnancy test following embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal females between the ages of 18 and 42 years
2. Body mass index (BMI) of 18-34
3. Early follicular phase (day 2-4) Follicle stimulating hormone (FSH) <15 IU/L and Estradiol (E2) within normal limits
4. Documented history of infertility (e.g., unable to conceive for at least one year, or for 6 months for women >38 years of age, or bilateral tubal occlusion or absence, or male factor but excluding severe male factor requiring invasive or surgical sperm retrieval. Donor sperm may be used.)
5. Transvaginal ultrasound at screening consistent with findings adequate for assisted reproductive technology (ART) with respect to uterus and adnexa
6. Signed informed consent

Exclusion Criteria:

1. Gestational or surrogate carrier, donor oocyte
2. Presence of any clinically relevant systemic disease (e.g., insulin-dependent diabetes mellitus, uterine cancer)
3. Surgical or medical condition which, in the judgment of the Investigator or Sponsor, may interfere with absorption, distribution, metabolism, or excretion of the drugs to be used
4. Previous In vitro fertilization (IVF) or Assisted reproductive technology (ART) failure due to a poor response to gonadotropins. Poor response is defined as development of 2 mature follicles or history of >2 previous failed in vitro fertilization (IVF) cycles.
5. History of recurrent pregnancy loss (>2).
6. Presence of abnormal uterine bleeding of undetermined origin
7. Current or recent substance abuse, including alcohol or smoking >10 cigarettes per day
8. Refusal or inability to comply with the requirements of the Protocol for any reason, including scheduled clinic visits and laboratory tests
9. Participation in any experimental drug study within 30 days prior to Screening
10. Severe male factor requiring invasive or surgical sperm retrieval (e.g., microsurgical epididymal sperm aspiration [MESA], testicular sperm extraction [TESE])

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (7):
- United States (7):
  - Huntington Reproductive Center, Pasadena, California
  - San Diego Fertility Center, San Diego, California
  - Conceptions Reproductive Associates of Colorado, Littleton, Colorado
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - The Advanced IVF Institute; Charles E. Miller, MD & Associates, Naperville, Illinois
  - A Woman's Center for Reproductive Medicine, Baton Rouge, Louisiana
  - Center for Assisted Reproduction, Bedford, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred ninety one (191) participants were screened from 6 study centers in the US; 173 of these participants were eligible for randomization. Six subjects did not receive their respected treatment and two subjects withdrew consent, 165 subjects were included in the statistical analyses
Groups:
- Menopur/Endometrin: Highly purified menotropin (Menopur®) 225 IU by subcutaneous injection once per day from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone vaginal insert (Endometrin®) 100 mg inserted vaginally 2 or 3 times daily (BID or TID) starts on the day following oocyte retrieval and continues for a total duration of 10 weeks or until a negative pregnancy test is obtained.
- Menopur/Progesterone in Oil: Highly purified menotropin 225 IU by subcutaneous injection once per day from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone in oil injections 50 mg by intramuscular injection (IM) once per day start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
- Follistim/Endometrin: Follitropin beta (Follistim®) 225 IU (up to 450 IU) by subcutaneous injection once per day from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone vaginal insert (Endometrin®) 100 mg inserted vaginally 2 or 3 times daily (BID or TID) starts on the day following oocyte retrieval and continues for a total duration of 10 weeks or until a negative pregnancy test is obtained.
- Follistim/Progesterone in Oil: Follitropin beta (Follistim®) 225 IU (up to 450 IU) by subcutaneous injection once per day from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone in oil injections 50 mg by intramuscular injection (IM) once per day start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
Period: Overall Study
Arm/Group | Menopur/Endometrin | Menopur/Progesterone in Oil | Follistim/Endometrin | Follistim/Progesterone in Oil
Started | 42 | 42 | 42 | 39
Completed | 18 | 16 | 17 | 17
Not Completed | 24 | 26 | 25 | 22
Not completed — Stimulation failure | 4 | 0 | 3 | 3
Not completed — Inadequate number of oocytes retrieved | 0 | 0 | 0 | 1
Not completed — Cycle cancelled | 0 | 1 | 1 | 1
Not completed — Risk of ovarian hyperstimulation syndrom | 0 | 0 | 0 | 1
Not completed — No positive serum pregnancy | 17 | 20 | 14 | 10
Not completed — Pregnancy not confirmed by ultrasound | 1 | 0 | 1 | 0
Not completed — Pregnancy loss/miscarriage | 0 | 2 | 0 | 3
Not completed — Other | 2 | 3 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menopur/Endometrin | Menopur/Progesterone in Oil | Follistim/Endometrin | Follistim/Progesterone in Oil | Total
Number analyzed (Participants) | 42 | 42 | 42 | 39 | 165
Age Continuous [Mean (Standard Deviation); unit: years] | 33.5 (4.1) | 33.2 (4.8) | 34.0 (4.3) | 33.9 (4.3) | 33.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 42 | 39 | 165
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 32 | 35 | 31 | 32 | 130
  African American | 5 | 1 | 2 | 2 | 10
  Asian | 4 | 2 | 6 | 2 | 14
  Hispanic | 1 | 4 | 3 | 1 | 9
  Other | 0 | 0 | 0 | 2 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (4.1) | 23.8 (3.0) | 25.0 (3.3) | 25.6 (4.5) | 24.6 (3.8)
Follicle-stimulating hormone level [Mean (Standard Deviation); unit: mIU/mL] | 7.4 (2.3) | 7.1 (2.2) | 6.9 (2.0) | 6.9 (2.9) | 7.3 (2.3)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Follicles Observed at Day 15
Description: The mean number of follicles observed in both ovaries at the last transvaginal ultrasound in the stimulation phase.
Time Frame: Day 15
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: follicles
Groups:
- Menopur: Highly purified menotropin (Menopur) 225 IU by subcutaneous injection once per day from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  This group combines the two treatment arms that use Menopur for ovarian stimulation. This treatment is followed by luteal support using either progesterone vaginal insert (Endometrin®) or progesterone in oil.
- Follistim: Follitropin beta (Follistim®) 225 IU by subcutaneous injection once per day from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  This group combines the two treatment arms that use Follistim for ovarian stimulation. This treatment is followed by luteal support using either progesterone vaginal insert (Endometrin®) or progesterone in oil.
Arm/Group | Menopur | Follistim
Number analyzed (Participants) | 84 | 81
follicles | 15.6 (8.6) | 16.2 (8.4)

2. Secondary Outcome: Number of Oocytes Retrieved at Day 18
Description: The mean number of oocytes retrieved within 34-36 hours of human chorionic gonadotropin (hCG) administration.
Time Frame: Approximately Day 18
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication and had oocytes retrieved.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Menopur | Follistim
Number analyzed (Participants) | 79 | 74
oocytes | 11.5 (6.3) | 13.8 (7.9)

3. Secondary Outcome: Proportion of Oocytes Fertilized of the Total Number of Oocytes Retrieved
Description: The proportion of the number of oocytes inseminated (fertilized) of the total number of oocytes retrieved.
Time Frame: Approximately Day 19
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: proportion of oocytes retrieved
Arm/Group | Menopur | Follistim
Number analyzed (Participants) | 79 | 73
proportion of oocytes retrieved | 0.3 (0.4) | 0.3 (0.4)

4. Secondary Outcome: Number of Embryos Transferred at Three Stages of Development
Description: The number of embryos, morula and blastocytes transferred to the study participant on either day 3 or day 5 following fertilization.
Time Frame: Approximately Day 24
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication and had embryos transferred.
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | Menopur | Follistim
Number analyzed (Participants) | 78 | 69
embryos
  Number of Embryos transferred | 2.1 (0.7) | 2.4 (0.7)
  Number of Morula transferred | 0.0 (0.1) | 0.1 (0.4)
  Number of Blastocytes transferred | 0.9 (1) | 0.9 (1)

5. Secondary Outcome: Number of Embryos Frozen at Day 24
Description: The number of embryos that were not transferred but instead were frozen for future use.
Time Frame: Approximately Day 24
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication and had oocytes fertilized
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | Menopur | Follistim
Number analyzed (Participants) | 78 | 69
embryos | 1.9 (2.9) | 1.6 (2.5)

6. Secondary Outcome: Participants With Cycle Cancellation Following One In Vitro Fertilization (IVF) Treatment Cycle
Description: A count of participants whose discontinuation was clearly documented on the study completion/termination form as 1) due to cycle cancelled or 2) cycle cancellation for risk of ovarian hyperstimulation syndrome (OHSS).
Time Frame: Day 1 to Day 24
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Menopur/Endometrin | Menopur/Progesterone in Oil | Follistim/Endometrin | Follistim/Progesterone in Oil
Number analyzed (Participants) | 42 | 42 | 42 | 39
participants | 0 | 1 | 1 | 2

7. Primary Outcome: Percentage of Participants With Ongoing Pregnancy at Week 8
Description: The ongoing pregnancy was defined as a positive fetal heart movement (motion) at approximately six weeks of gestation and confirmed in a follow-up pregnancy ultrasound.
Time Frame: Week 8 (Week 6 of gestation)
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Menopur/Endometrin | Menopur/Progesterone in Oil | Follistim/Endometrin | Follistim/Progesterone in Oil
Number analyzed (Participants) | 42 | 42 | 42 | 39
percentage of participants | 45.2 | 45.2 | 42.9 | 48.7

8. Secondary Outcome: Participants With Biochemical Pregnancy at Day 38
Description: Biochemical pregnancy is a positive β-hCG pregnancy test 12-14 days post embryo transfer.
Time Frame: approximately day 38 (Day 14 post embryo transfer)
Population: Intent-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication and had an embryo transfer
Measure: Number; unit: participants
Arm/Group | Menopur/Endometrin | Menopur/Progesterone in Oil | Follistim/Endometrin | Follistim/Progesterone in Oil
Number analyzed (Participants) | 38 | 40 | 36 | 33
participants | 21 | 20 | 22 | 23

9. Secondary Outcome: Participants With Clinical Pregnancy at Week 7
Description: Clinical pregnancy is the confirmation of the presence of intrauterine gestational sacs on pregnancy ultrasound examination.
Time Frame: approximately week 7
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Menopur/Endometrin | Menopur/Progesterone in Oil | Follistim/Endometrin | Follistim/Progesterone in Oil
Number analyzed (Participants) | 38 | 40 | 36 | 33
participants | 19 | 19 | 18 | 20

10. Secondary Outcome: Participants With Adverse Events (AEs), Including Ovarian Hyperstimulation Syndrome (OHSS)
Description: Number of participants with adverse events (AEs) that started after first treatment. Severity used a three point scale:
  mild=awareness of signs/symptoms, but no disruption of usual activity moderate=event sufficient to affect usual activity (disturbing) severe=event causes inability to work or perform usual activities (unacceptable)
  Relatedness to study treatment used a four point scale: unrelated, unlikely, possible, probable.
  Seriousness refers to death, hospitalization, a life-threatening experience, persistent or significant disability/incapacity, or congenital anomaly.
Time Frame: Day 1 - week 12
Population: Safety population all randomized and treated participants. The safety population is identical intent-to- treat (ITT) population in this study
Measure: Number; unit: participants
Arm/Group | Menopur/Endometrin | Menopur/Progesterone in Oil | Follistim/Endometrin | Follistim/Progesterone in Oil
Number analyzed (Participants) | 42 | 42 | 42 | 39
participants
  With at least one adverse event | 20 | 18 | 18 | 21
  Mild or moderate adverse event | 20 | 18 | 18 | 21
  Severe adverse event | 1 | 0 | 2 | 0
  Serious adverse event | 0 | 1 | 1 | 0
  Unrelated or unlikely adverse event | 15 | 13 | 17 | 14
  Possibly or probably related adverse event | 10 | 8 | 7 | 15

11. Secondary Outcome: Number of Live Births
Time Frame: Approximately 10 months
Population: Database was locked prior to all participants giving birth.
Measure: Number; unit: live births
Arm/Group | Menopur/Endometrin | Menopur/Progesterone in Oil | Follistim/Endometrin | Follistim/Progesterone in Oil
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from Day 1 to Week 12.
Description: Multiple events in the same system organ class for a subject are only counted once for that system organ class.
Arm/Group | Menopur/Endometrin | Menopur/Progesterone in Oil | Follistim/Endometrin | Follistim/Progesterone in Oil
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/42 | 1/42 | 0/39
Other Adverse Events (participants affected / at risk) | 20/42 | 18/42 | 18/42 | 21/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menopur/Endometrin (N=42) | Menopur/Progesterone in Oil (N=42) | Follistim/Endometrin (N=42) | Follistim/Progesterone in Oil (N=39)
Ovarian hyperstimulation syndrome with ascites (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Hyperemesis gravidarum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menopur/Endometrin (N=42) | Menopur/Progesterone in Oil (N=42) | Follistim/Endometrin (N=42) | Follistim/Progesterone in Oil (N=39)
Abdominal distension (Gastrointestinal disorders) | 4 | 6 | 3 | 5
Abdominal pain lower (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 5 | 3 | 8
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3 | 5 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2
Adnexa uteri pain (Reproductive system and breast disorders) | 6 | 7 | 6 | 9
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 3 | 1 | 1 | 8
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Injection site discomfort (General disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site oedema (General disorders) | 0 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 0 | 0 | 1
Irritability (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 2 | 1 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injection site anaesthesia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0
Bladder pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1 | 1
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine spasm (Reproductive system and breast disorders) | 1 | 1 | 2 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This was an exploratory study that could be used as the basis for larger, adequately-powered studies. This limitation is the reason no statistical analyses are offered for study outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor.

Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.